CLINICAL TRIAL: NCT01233635
Title: Secondary Prevention of Atrial Fibrillation (Impact of Renin-Angiotensin-Aldosterone System Inhibition)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: inadequate enrollment rate
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0507061
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2016-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

ARMS (3):
- A Group 1 no drug (Experimental): Patients who have not taken ACE/ARB, randomized to no drug.
  Interventions: Other: no drug
- A Group 2 (Experimental): Patients who have not taken ACE/ARB, randomized to take cozaar.
  Interventions: Drug: start cozaar
- B (Experimental): Patients currently taking ACE/ARB will have their prescription changed to cozaar.
  Interventions: Drug: continue cozaar

INTERVENTIONS:
Other: no drug — none, no drug
  Arms: A Group 1 no drug
Drug: start cozaar — start cozaar
  Arms: A Group 2
Drug: continue cozaar — continue cozaar
  Arms: B

SUMMARY:
In the present application, we propose to refine and extend current insight into AAF mechanism and therapy by examining the importance of pharmacologic RAAS inhibition, ACE genotype, and their interaction in secondary AF prevention. We have 3 specific aims:

1. To confirm that RAAS inhibition therapy reduces the incidence of AF recurrence.
2. To test the hypothesis that the incidence of AF recurrence in the absence of RAAS inhibition therapy is higher among patients with the D allele.
3. To explore the hypothesis that RAAS inhibition therapy is more effective for preventing AF recurrence in patients with the DD genotype than in those with DI or II genotypes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be in atrial fibrillation confirmed by 12 lead EKG.
* blood pressure > 90 mmHg
* Patient without cardiopulmonary symptoms
* 18+ years of age

Exclusion Criteria:

* Contraindiction to warfarin
* Recent (within 6 months) MI or cardiac revascularization
* Recent (within 6 months) CVA or TIA
* NYHA Class IV CHF
* Active thyroid disease
* Major hepatic dysfunction
* Renal dysfunction (>2 mg/dL)
* Hyperkalemia (>4.6 mEq/L)
* Hyponatremia (<130 mEq/L)
* Currently taking a Vaughn-Williams Type I or III antiarrhythmic drug
* History of ARB intolerance
* Contraindication to ARB therapy
* Pregnancy
* Female of childbearing age
* Age < 18 years of age
* Inability to give informed consent
* Other medical conditions calling 1 year survival into question

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2005-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
AF burden | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC CVI, Pittsburgh, Pennsylvania, United States